CLINICAL TRIAL: NCT01267981
Title: Impact of Small Bowel Preparation Using Polyethylene Glycol for Endoscopic Video-capsule (EVC)Exploration in Unexplained Gastrointestinal Bleedings
Brief Title: Efficacy of Small Bowel Preparation in Capsule Endoscopy
Acronym: PREPINTEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RB 09.091
Record Dates: First submitted 2010-12-27; First posted 2010-12-29 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2017-11

CONDITIONS: Gastrointestinal Bleedings
Keywords: Small bowel; video-capsule endoscopy; gastrointestinal bleeding; polyethylene glycol
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Preparation 1 (Placebo Comparator): Standard diet: the day before video-capsule exploration : Drink only clears liquids after the lunch, fasting from 22 hours except usual drugs with a mouthful water.
  Interventions: Drug: Standard diet
- Preparation 2 (Active Comparator): Standard diet : the day before video-capsule exploration : Drink only clears liquids after the lunch, fasting from 22 hours except usual drugs with a mouthful water.
  500 ml of polyethylene glycol 30 minutes after the ingestion of video-capsule endoscopy.
  Interventions: Drug: Standard Diet + 500 ml of polyethyleneglycol
- Preparation 3 (Active Comparator): Standard diet : the day before video-capsule exploration : Drink only clears liquids after the lunch, fasting from 22 hours except usual drugs with a mouthful water.
  2 liters of polyethylene glycol between 7 pm and 9 pm.
  500 ml of polyethylene glycol, 30 minutes after the ingestion of video-capsule endoscopy.
  Interventions: Drug: Standard diet + 2 liters of polyethylene glycol the day before + 500ml of polyethylene glycol

INTERVENTIONS:
Drug: Standard diet — After the lunch the day before the exploration, drink only clear liquids and stop solid food.
  From 10 pm, stay fasting, don't drink except the usual drugs taken with mouthful of water until the exploration by video-capsule endoscopy.
  Arms: Preparation 1
Drug: Standard Diet + 500 ml of polyethyleneglycol — Apply the standard diet and drink 500 ml of polyethylene glycol 30 minutes after the endoscopy video-capsule ingestion.
  Arms: Preparation 2
Drug: Standard diet + 2 liters of polyethylene glycol the day before + 500ml of polyethylene glycol — apply the standard diet and drink 2 liters of polyethylene glycol between 19h and 21h the day before exploration. Then drink 500 ml of polyethylene glycol 30 minutes after the endoscopy video-capsule ingestion.
  Arms: Preparation 3

SUMMARY:
The best preparation of small bowel is still unknown. The primary aim of this study is to evaluate the polyethylene glycol (PEG) impact of small bowel preparation for unexplained gastrointestinal bleeding exploration. Three different preparations are evaluated in this study.

DETAILED DESCRIPTION:
Now days, the endoscopic video-capsule is the more appropriate exam for unexplained gastrointestinal bleeding exploration. The responsible damage of this unexplained bleeding are frequently small vascular damages, hard to be detected in the bowel or ulcerations or tumors. The exam quality can be limited by food residues, bubbles or bile.

30% of damage are probably undetectable because of a lack of visibility. An efficient preparation will probably increased the quality of the video-capsule exploration.

The bowel exploration by endoscopy video-capsule will be realized in the usual condition. The study included 4 steps:

1. Inclusion
2. Randomization
3. Video-capsule exploration
4. Reading of the video-capsule exam by endoscopist doctors who are in blind.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old.
* Patients who have an indication for video-capsule endoscopy exploration for unexplained gastrointestinal bleeding associated with anaemia (man : haemoglobin <13 g/dl and woman haemoglobin <12g/dl)
* Less than one year Endoscopic assessment by colonoscopy and gastroscopy
* Not participated to an another clinic study.
* Written consent.

Exclusion Criteria:

* Age<18 years old.
* General physical health deterioration such as dehydration or cardiac insufficiency.
* Clinical or radiological suspicion of digestive stenosis.
* Oral iron taking in the 4 days before video-capsule exploration.
* Functional or organic disorders of the gulp
* Pregnant women.
* Sensibility known about the polyethylene glycol.
* No signed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2010-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Compare the frequencies of the diagnoses of clinically significant lesions | at the end of video-capsule exploration
  Compare the frequencies of the diagnoses of clinically significant lesions (P1 or P2)obtained with and without polyethylene glycol preparation for patients investigated by video-capsule endoscopy who have an unexplained digestive bleeding.

SECONDARY OUTCOMES:
The quality of the preparation and visibility of the bowel | at the end of video-capsule exploration
  Demonstrate an improvement in preparation quality and bowel visibility in the various segments of small bowel examined by video-capsule endoscopy
The clinical tolerance | 8 days after video-capsule exploration
  Evaluate the clinical tolerance and the acceptability of the bowel preparation with oral polyethylene glycol solution
The number of all the observed lesions | at the end of video-capsule exploration
  Estimate the number of all the observed lesions on the recording according to their hemorrhagic potential.
Compare different times | at the end of video-capsule exploration
  Compare gastric emptying time, the bowel transit time and the percentage complete medical exploration of small bowel for every group of patients (ileo- cecal valve exceeded).
Crossing (yes or no) of ileo-cecal valve by the EVC | At the end of video-capsule exploration

CONTACTS AND LOCATIONS:
Overall Officials: Franck CHOLET, MD, Principal Investigator — CHRU Brest
Locations (17):
- France (17):
  - Centre Hospitalier d'Avignon, Avignon
  - Cabinet privé, Béziers
  - Centre Hospitalier d'Avicenne, Bobigny
  - CHOLET, Brest
  - CHRU de Lille, Lille
  - Saint Philibert Hospital, Lomme
  - CH Bretagne Sud, Lorient
  - Edouard Herriot Hospital, Lyon
  - Hôpital de La Conception, Marseille
  - Hôpital de la Timone, Marseille
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital Cochin, Paris
  - Höpital Européen Geores Pompidou, Paris
  - CH de Cornouaille Quimper, Quimper
  - Centre Hospitalier de Saint Brieuc, Saint-Brieuc
  - Hôpital Privé de L'Est Lyonnais, Saint-Priest
  - CH Bretagne Atlantique, Vannes

REFERENCES:
- [Derived] Rahmi G, Cholet F, Gaudric M, Filippi J, Duburque C, Bramli S, Quentin V, Alavi Z, Nowak E, Saurin JC, Cellier C, Queneherve L; PREPINTEST working group. Effect of Different Modalities of Purgative Preparation on the Diagnostic Yield of Small Bowel Capsule for the Exploration of Suspected Small Bowel Bleeding: A Multicenter Randomized Controlled Trial. Am J Gastroenterol. 2022 Feb 1;117(2):327-335. doi: 10.14309/ajg.0000000000001597. PMID 35041627